CLINICAL TRIAL: NCT01763112
Title: Influence of Training With Whole Body Vibration Device (Galileo) on Quality of Life (QoL), Exercise Capacity, as Well as on the Effects of Muscle Power and Muscle Function in Patients With Pulmonal Arterial Hypertension (PAH). (GALILEO PAH)
Brief Title: Training With Whole Body Vibration Device in Patients With PAH
Acronym: GALILEO-PAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klinikum der Universität Köln (Other)
Responsible Party: Principal Investigator, Felix Gerhardt, PhD, Klinikum der Universität Köln
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Artery Hypertension
Keywords: Influence of training with whole body vibration device
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): This group will not do any specific training baseline and week 4 investigation will be done only
- Exercise Group Galileo PAH (Active Comparator): The intervention/exercise group will do whole body vibration training on 4 days a week for 60 minutes over 4 weeks
  Interventions: Device: Exercise Group Galileo PAH

INTERVENTIONS:
Device: Exercise Group Galileo PAH — The intervention/exercise group will do whole body vibration training on 4 days a week for 60 minutes over 4 weeks
  Arms: Exercise Group Galileo PAH

SUMMARY:
Title of study / project: Influence of training with whole body vibration device on Quality of Life (QoL), exercise capacity, as well as on the effects of muscle power and muscle function in patients with pulmonal arterial hypertension (PAH). Background and rationale for the proposal:Capacity and the ability to exercise, in patients with PAH is limited. There is a few investigations evaluating the effects of the training with whole body vibration (wbv) in adults. It was shown that wbv-training could improve muscle power, QoL, body balance and had positive effects on the neuromuscular system. Primary scientific question addressed:Changes in muscle power, changes in 6-Minute Walk Distance (6MWD) and changes in QoL are to be evaluated.

DETAILED DESCRIPTION:
Study Design: Open Monocentric prospective randomized observational trial Study arms: Treatment group (4-weeks wbv training) planned 20 patients Control group: planned 20 patients Endpoint (-s): Changes in muscle power, changes in 6-Minute Walk Distance (6MWD), changes in QoL changes in peak VO2 (bike exercise test)

Major study procedures:

Blood samples, vital parameters, questionnaires, echocardiography, lung function test, blood gas analysis, bike exercise test, 6-Minute Walk test, ECG, Chair rising test, power plate measurement, walk across test

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-90 years
* Signed informed consent
* Symptomatic PAH (idiopathic, hereditary or associated with systemic scleroderma)
* Invasively confirmed PAH
* 6MWT ≥ 50 m
* Stable specific therapy for at least 2 months
* Ability to perform bike test
* Ability to perform wbv training
* NYHA/WHO-FC II-III

Exclusion Criteria:

* any other PAH/PH than idiopathic, hereditary or associated with systemic scleroderma
* Rehabilitation or other training concept performed within 2 months before inclusion
* pregnancy
* acute thrombosis
* newly implanted Hip or Knee
* recent bone fracture
* Disability to confirm consent
* NYHA/WHO-FC IV

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
changes in 6-Minute Walk Distance (6MWD) | baseline and week 4

SECONDARY OUTCOMES:
Changes in Quality of life | baseline and week 4
Changes in peak Vo2 | baseline and week 4
Changes in muscle power | baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Felix Gerhardt, PhD, Principal Investigator — Klinik III für Innere Medizin Uniklinik Köln; Stephan Rosenkranz, PhD, Principal Investigator — Klinik III für Innere Medizin der Uniklinik Köln
Locations (1):
- Spezialambulanz für pulmonale Hypertonie Uniklinik Köln, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Gerhardt F, Dumitrescu D, Gartner C, Beccard R, Viethen T, Kramer T, Baldus S, Hellmich M, Schonau E, Rosenkranz S. Oscillatory whole-body vibration improves exercise capacity and physical performance in pulmonary arterial hypertension: a randomised clinical study. Heart. 2017 Apr;103(8):592-598. doi: 10.1136/heartjnl-2016-309852. Epub 2017 Jan 18. PMID 28100544